CLINICAL TRIAL: NCT03955887
Title: Mitochondrial Dysfunction of Alveolar and Circulating Immune Cells During Acute Respiratory Distress Syndrome: Impact of Infectious Aggression and Alveolar Stretching as a Result of Mechanical Ventilation.
Acronym: PNEUMOCHONDRIE
Status: Terminated | Type: Observational
Why Stopped: technical difficulties
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BLOT MSD-APJ 2018
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Lung Diseases; Mechanical Ventilation; Bronchoalveolar Lavage
MeSH Terms: conditions — Lung Diseases | interventions — Bronchoalveolar Lavage Fluid; Venous Pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchialveolar lavage fluid (10 mL) Venous blood (12 mL)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: Patients with severe acute lung disease requiring mechanical ventilation
  Interventions: Biological: bronchoalveolar lavage fluid (BAL); Biological: Venous blood
- Control: Patients receiving routine bronchoalveolar lavage for a pathology not suspected of acute infection
  Interventions: Biological: bronchoalveolar lavage fluid (BAL); Biological: Venous blood

INTERVENTIONS:
Biological: bronchoalveolar lavage fluid (BAL) — Recovery of a 10 mL volume of BAL fluid, performed as part of patient care
Biological: Venous blood — Collection of 3 additional blood tubes (12 ml) during a blood sample taken as part of patient care

SUMMARY:
Sepsis leads to a deregulated host response that can lead to organ failure. During sepsis, experimental and clinical data suggest the occurrence of mitochondrial dysfunctions, particularly in circulating muscle and monocytes, which may contribute to organ failure and death.

Lower respiratory infection is the leading cause of death from infectious causes. Mechanical ventilation (MV) is required in 20% of cases of bacterial pneumopathy with Streptococcus pneumoniae (S.p.) , with mortality reaching 50%. There are then frequently criteria for acute respiratory distress syndrome (ARDS), combining bilateral lung involvement and marked hypoxemia.

Cyclic stretching of lung cells induced by MV causes sterile inflammation and tissue damage (i.e. ventilator-induced lung injury [VILI]), which can cause cellular dysfunction that alter the immune response, particularly during ARDS. This is why the application of a so-called protective MV is then required. However, this does not prevent about one-third of patients from showing signs of alveolar overdistension, as evidenced by an increase in motor pressure (MP) (MP≥ 15 cmH2O), associated with an increase in mortality.

The deleterious effects of MV could be explained by the occurrence of mitochondrial abnormalities. Indeed, the cyclic stretching of lung cells leads to dysfunction in the respiratory chain and the production of free oxygen radicals (FOS), altering membrane permeability. These phenomena could promote VILI, facilitate the translocation of bacteria from the lung to the systemic compartment and lead to alterations in immune response.

In our model of S.p. pneumopathy in rabbits, animals on MV develop more severe lung disorders (lack of pulmonary clearance of bacteria, bacterial translocation in the blood, excess mortality), compared to animals on spontaneous ventilation (SV). Intracellular pulmonary mitochondrial DNA (mtDNA) concentrations, a reflection of the mitochondrial pool, are significantly decreased in ventilated rabbits compared to SV rabbits and in infected rabbits compared to uninfected rabbits. At the same time, the mitochondrial content of circulating cells decreased early (H8) in all infected rabbits, but was only restored in rabbits in SV, those who survived pneumonia (Blot et al, poster ECCMID 2015, submitted article). These data suggest an alteration in the mechanisms that restore mitochondrial homeostasis (mitochondrial biogenesis and mitophagy) during the dual infection/MV agression, which may explain the observed excess mortality. Other work by our team illustrates the importance of these phenomena by showing in a mouse model of polymicrobial infection that inhibition of mitophagia in macrophages promotes survival (Patoli et al, in preparation). Human data on this subject are non-existent.

The phenomena of mitochondrial dysfunction nevertheless deserve to be explored in humans during the combined MV/pneumopathy aggression in order to understand its possible impact on the effectiveness of the host's immune response. In a personalized medicine approach, these data would open up prospects for targeted therapies, capable of activating mitochondrial biogenesis and/or modulating mitophagia, to prevent organ dysfunction and mortality during severe CALs treated with antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has given his non-opposition (or non-opposition obtained from close relative of ventilated patients, who will be informed as soon as possible).
* Adult patient
* Group 1: patient with:

  * Acute pneumonitis defined by: Signs and acute symptoms of pneumonia (new or worsening within the last 7 days), at least 2 of which are:

    * Coughing
    * Purulent sputum
    * Dyspnea
    * Chest pain
    * Temperature < 35°C or ≥ 38°C And a new pulmonary radiological infiltrate (x-ray or CT scan on admission)
  * Not acquired under mechanical ventilation
  * Complicated from ARDS according to the new Berlin definition, Chest x-ray finding bilateral parenchymal opacities not fully explained by pleural effusions, nodules or atelectasis. Respiratory distress not explained by cardiac dysfunction or overfilling. An echocardiogram will be performed in case of diagnostic uncertainty. PaO2/FiO2 report < 300 and PEP ≥ 5 cmH2O
  * Requiring the use of MV.
  * With a diagnostic BAL performed within 72 hours of the start of the MV
* Group 2: Patients:

  * No fever during the last 15 days (reported or measured ≥ 37.8°C).
  * Not under MV,
  * Undergoing BAL for a reason other than acute infection (e.g. chronic interstitial syndrome, nodule or lung mass).

Exclusion Criteria:

* Patient not affiliated to the national health insurance system
* Major under judicial protection
* Pregnant, parturient or breastfeeding woman
* Known primary or secondary immune deficiency (radiotherapy, chemotherapy, immunosuppressive therapy or systemic corticosteroid therapy (>10mg/day prednisone equivalent for more than 7 days) within 6 months before inclusion, HIV infection, primary cellular immune deficiency)
* Patients with treatment known to modulate mitochondrial function, biogenesis and/or mitophagia (chloroquine, hydroxychloroquine, rapamycin, carbamazepine, resveratrol, metformin, sildenafil)
* Patients with pulmonary fibrosis or cystic fibrosis known to be associated with mitochondrial alterations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admited in the Intensive Care Unit and the Pneumology Intensive Care Unit of the CHU Dijon Bourgogne
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
Active mitochondria content of alveolar macrophages | Through study completion, an average of 19 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

REFERENCES:
- [Result] Blot M, Bour JB, Quenot JP, Bourredjem A, Nguyen M, Guy J, Monier S, Georges M, Large A, Dargent A, Guilhem A, Mouries-Martin S, Barben J, Bouhemad B, Charles PE, Chavanet P, Binquet C, Piroth L; LYMPHONIE study group. The dysregulated innate immune response in severe COVID-19 pneumonia that could drive poorer outcome. J Transl Med. 2020 Dec 3;18(1):457. doi: 10.1186/s12967-020-02646-9. PMID 33272291
- [Derived] Blot M, Jacquier M, Aho Glele LS, Beltramo G, Nguyen M, Bonniaud P, Prin S, Andreu P, Bouhemad B, Bour JB, Binquet C, Piroth L, Pais de Barros JP, Masson D, Quenot JP, Charles PE; Pneumochondrie study group. CXCL10 could drive longer duration of mechanical ventilation during COVID-19 ARDS. Crit Care. 2020 Nov 2;24(1):632. doi: 10.1186/s13054-020-03328-0. PMID 33138839